CLINICAL TRIAL: NCT04932174
Title: Effect of High Intensity Interval Training Versus Low Intensity Continuous Training on Physical Fitness Among Overweight Adult
Brief Title: High Intensity Interval Training Versus Low-intensity Continuous Training on Physical Fitness Among Overweight Adult
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Heba Yasser, Principal Investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hebayasser_MSc
Record Dates: First submitted 2021-06-13; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Overweight; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity Interval Training (Experimental): Group 2: the included 15 subjects will participate in High intensity Interval training exercise running on treadmill for 12 weeks, 3 times / week.
  Interventions: Other: High-intensity Interval Training
- Low-intensity Continuous Training (Active Comparator): Group 1: the included 15 subjects will participate in low intensity continuous exercise on treadmill for 12 weeks, 3 times / week
  Interventions: Other: Low-intensity Continuous Training

INTERVENTIONS:
Other: High-intensity Interval Training — Consisting of the following program:
  * Warming up period for 10 minutes at 60-70% of HR max.
  * Training phase 4x4 min intervals at 85-90% of HRmax with a 3 min active recovery at 70% of HRmax between each interval.
  * Duration of HIIT 4 minute
  * Number of interval per session 4
  * Duration of rest interval 3 minute 3-10 min cool-down period, giving a total of 60 min.
  Arms: High-intensity Interval Training
Other: Low-intensity Continuous Training — Consisting of the following program:
  * Warming up period for 10 minutes.
  * Training phase for 60-minute walking on a treadmill at intensity 40-50% HRR (1- 6) weeks then 60-70% HRR (7-12) weeks.
  * cooling down period for 10 minutes.
  Arms: Low-intensity Continuous Training

SUMMARY:
The purpose of the study is to compare the effect of high intensity interval training and low intensity training on physical fitness among adult overweight.

DETAILED DESCRIPTION:
Excess body weight has been shown to negatively influence musculoskeletal health and may limit physical function. Thus, there is a need for effective interventions to reduce body weight in those individuals who may already be overweight or obese. Physical activity can be an important component of lifestyle interventions for weight loss. Thus, it is important for clinicians, health care providers, and health-fitness professionals to recognize the influence of physical activity on body weight and to understand recommendations that can affect physical activity behavior. Several studies reported that HIIT can improve cardiorespiratory fitness (increase vo2 max) in adults with varied body weight and health status.

High intensity interval training induced improvements in insulin sensitivity, blood pressure, and body composition more consistently occur in adults with overweight, with or without high risk of cardiovascular disease and diabetes especially if these participate in prolonged exercise program up to 12 or more weeks.

Low intensity exercise has been shown to have a range of physiological and biochemical effects during a subsequent bout of exercise Low intensity exercise would result in muscle acetyl group accumulation and thereby would accelerate mitochondrial ATP production (and reduce ATP production from nonoxidative routes) during a subsequent bout of moderate intensity exercise. In accordance with these changes, we also hypothesized that the vo2 on-kinetics during moderate intensity exercise would be accelerated when preceded by low intensity exercise .

The significant behind this study came up with the importance to declare the effect of high intensity interval training on improving physical fitness and body composition which be more suitable for overweight active people that don't have time to practice prolonged exercise during the week and this study also will investigates the effect of low intensity exercise on physical fitness and body composition to declare where is going to be beneficial for overweight sedentary subjects and compare it is effect with pervious.

This study will be designed to provide a guideline about the effect of high intensity interval training& low intensity training exercise on physical fitness in the overweight adult patient.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) will be ≥ 25 -29.9 kg/m².
2. Age will be ranging from 20 to 30 years.
3. Waist circumference >88cm2 in men and >102cm2 in women.
4. Content of body fat will be assisted by electrical bioimpedence≥33%.
5. Stable body weight in the month prior to the trial.
6. Follow instructions for healthy life style.

Exclusion Criteria:

1. Patients with musculoskeletal deformities and disorders.
2. Patients with other neuromuscular disorders.
3. Patients with foot deformities and ulcers.
4. Patients with lower limb operations.
5. Smoking cigarettes, thyroid diseases.
6. History of coronary artery disease Asthma, chronic obstructive pulmonary diseases.
7. poorly controlled hypertension (mean systolic blood pressure (SBP) > 140 mm Hg and/or mean diastolic blood pressure (DBP) > 90 mm Hg) during the month prior to the trial.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in body Weight | Baseline and 2 months post-intervention
  Assessment via using body weight scale with height (m) scale to be able to calculate body mass index (Kg) to all subjects before starting the study BMI= Weight (KG) /Height2 (M2)
Assessing the change in Waist hip ratio | Baseline and 2 months post-intervention
  Assessment via using was measured to the nearest 0.1 cm by using a flexible steel tape at the level of umbilicus, and hip circumference (HC) was measured at the widest level over the greater trochanters.
Assessing the change in body fat | Baseline and 2 months post-intervention
  Assessment through bioelectrical impedance analysis by using a Body Composition Analyzer (TANITA Corporation, Japan).
Assessing the change Cardiorespiratory fitness | Baseline and 2 months post-intervention
  Assessment via using Shuttle run test The 20-m shuttle run (20MSR) test, also called the ''Course Navette'', "PACER", or "Multistage fitness test", is probably the most widely used field test for estimating cardiorespiratory fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Yasser, Demonstrator, Principal Investigator — Horus University in Egypt
Locations (1):
- Outpatient clinic - Faculty of Physical Therapy - Horus University, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No